CLINICAL TRIAL: NCT02400840
Title: Acute Heart Graft Rejection Screening by Cardiac Magnetic Resonance Imaging
Acronym: DRAGON
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not feasable yet, due to evolution in the patients' care
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2013/153/HP
Record Dates: First submitted 2015-01-26; First posted 2015-03-27 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart graft rejection (Experimental): Assessment of cardiac allograft recipient with rejection by Cardiac MRI with gadobenic acid intravenous injection 0.2 ml/kg one time
  Interventions: Procedure: cardiac MRI; Drug: gadobenic acid intravenous injection 0.2 ml/kg
- No rejection (Active Comparator): Assessment of cardiac allograft recipient without any rejection by Cardiac MRI with gadobenic acid intravenous injection 0.2 ml/kg one time
  Interventions: Procedure: cardiac MRI; Drug: gadobenic acid intravenous injection 0.2 ml/kg

INTERVENTIONS:
Procedure: cardiac MRI — Cardiac MRI is done using gadobenic acid intravenous injection 0.2 ml/kg one time
Drug: gadobenic acid intravenous injection 0.2 ml/kg — gadobenic acid intravenous injection 0.2 ml/kg is used one time for cardiac MRI assessment

SUMMARY:
Acute heart allograft rejection is a common complication after orthotopic heart transplantation. Primary objective of this study is to assess cardiac MRI as a tool for acute heart graft rejection screening, by detecting changes in myocardium structure especially extracellular volume.

DETAILED DESCRIPTION:
Acute heart allograft rejection is a common complication after orthotopic heart transplantation. It can lead to multiple cardiac injuries and sometimes to patient's death. Currently, acute heart graft rejection screening is based on invasive strategies. Gold standard is represented by endomyocardial biopsies which provide side effects risk, rare but potentially fatal for the recipient. Cardiac MRI is an imaging tool recently used in cardiology. It is a non-invasive without any X-Ray exposition method well adapted to assess cardiac function and cardiac muscle composition. Cardiac MRI is probably a great tool to help the screening of acute heart allograft rejection, by detecting changes in myocardium structure. MRI validation as a screening tool for heart allograft rejection detection could help to reduce endomyocardial biopsies realised after orthotopic heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Orthotopic heart transplantation patients
* Endomyocardial biopsies < 72h
* Estimated glomerular filtration ratio >30ml/min (calculated by Cockcroft formula for patients age < 65 yo or MDRD for patients age >65 ans)
* Patients affiliated to French national health insurance
* For pre-menopausal female patients, negative pregnancy test
* Patient's consent form signature
* Patient with correct French writing and speaking comprehension

Exclusion Criteria:

* Endomyocardial biopsies showing acute cellular rejection grade 1R or antibodies mediated rejection pAMR1
* Patient in need of renal dialysis
* Past history of allergic reaction or side effects after gadolinium infusion
* Hemodynamical instability
* MRI contra-indication (claustrophobia, ocular metallic objects, non MRI compatible cardiac device, neurological non RMI compatible device, osteosynthesis prosthesis older than 1980)
* Pregnant or breast feeding woman
* Patient participating to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Number of patient with an acute rejection detected using Cardiac MRI after orthotopic heart transplantation | Day 1

SECONDARY OUTCOMES:
Extracellular volume as measured by Cardiac MRI | Day 1
T1 as measured by Cardiac MRI | Day 1
T2 as measured by Cardiac MRI | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud GAY, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France